CLINICAL TRIAL: NCT05598138
Title: Clinical and Biological Strokes Collection in Reunion Island
Acronym: CoBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/CHU/40
Record Dates: First submitted 2022-10-19; First posted 2022-10-28 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): A blood sample (10 ml) will be taken for each patient included in the study
  Interventions: Biological: Biological Collection

INTERVENTIONS:
Biological: Biological Collection — A blood sample (10 ml) will be taken for each patient included in the study.

SUMMARY:
Cross-sectional regional multicenter hospital study of all neurological events (stroke, AIT and mimics) for diagnostic and prognostic purposes. Cost of illness study.

ELIGIBILITY:
Inclusion Criteria:

* affiliated to a social security scheme
* clinical signs suggestive of stroke : hemiparesis or hemiplegia, unilateral sensory disorder, language disorder, balance disorder, dizziness, loss of total or partial bilateral or monocular vision, sudden neurological deficit

Exclusion Criteria:

* current pregnancy
* Recent clinical history of head trauma
* patients aged < 18 years old
* patient under guardianship or curatorship
* Person deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
clinico-biological score | 24 hours after the stroke
  area under the diagnostic score curve identifying ischemic stroke, stroke hemorrhagic or mimics.

CONTACTS AND LOCATIONS:
Locations (2):
- Reunion (2):
  - CHU de La Réunion, Saint-Denis
  - CHU de La Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No